CLINICAL TRIAL: NCT06893302
Title: Bone Marrow Aspirate Injections in Knee Arthroscopy: A Randomized, Single-Blind, Controlled Trial
Brief Title: Impact of Bone-Marrow Aspirate Injections in Knee Arthroscopy
Acronym: BMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-2344
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-03

CONDITIONS: Chondral Lesion of the Knee; Meniscal Injuries; Cartilage Defects of the Knee; Osteoarthritis (OA) of the Knee
Keywords: knee arthroscopy; meniscal injury; knee debridement; meniscectomy; osteoarthritis; cartilage defect; chondral lesion; bone marrow aspirate; BMA
MeSH Terms: conditions — Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to receive arthroscopic debridement surgery with saline injection or arthroscopic debridement surgery supplemented with bone marrow aspirate (BMA) injection.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arthroscopic Debridement Surgery + Saline (Active Comparator): Arthroscopic debridement surgery is standard of care to treat the conditions that are within the inclusion criteria of the study, therefore it serves as an Active Comparator to the experimental arm which is the same procedure but with the addition of bone marrow aspirate (BMA) injection.
  Interventions: Procedure: Arthroscopic Debridement Surgery; Other: Saline
- Arthroscopic Debridement Surgery + Bone Marrow Aspirate (BMA) (Experimental): Arthroscopic debridement surgery is standard of care to treat the conditions that are within the inclusion criteria of the study. The study investigates the effect of combining the standard of care with a bone marrow aspirate (BMA), therefore this serves as the Active Experimental arm.
  Interventions: Biological: Bone Marrow Aspirate (BMA); Procedure: Arthroscopic Debridement Surgery

INTERVENTIONS:
Biological: Bone Marrow Aspirate (BMA) — Bone marrow aspirate (BMA) is being investigated as an augmentation to arthroscopic debridement surgery of the knee to treat conditions such as meniscal injuries, chondral defects, and low-grade osteoarthritis.
  Arms: Arthroscopic Debridement Surgery + Bone Marrow Aspirate (BMA)
Procedure: Arthroscopic Debridement Surgery — Arthroscopic debridement surgery of the knee is performed to treat conditions such as meniscal injuries, chondral defects, and low-grade osteoarthritis.
Other: Saline — Patients in the control arm of the study will receive arthroscopic debridement surgery along with a saline injection. This will be compared to the experimental arm, in which patients will receive arthroscopic debridement surgery along with a bone marrow aspirate injection.
  Arms: Arthroscopic Debridement Surgery + Saline

SUMMARY:
This study will examine whether using bone marrow aspirate (BMA) during knee arthroscopy surgery can improve patient outcomes. The investigators will enroll 50 patients who need knee arthroscopy surgery for meniscus injuries or cartilage damage. Like flipping a coin, patients will be randomly assigned to one of two groups of 25 patients each. One group will receive standard arthroscopic surgery plus an injection of bone marrow aspirate, while the other group will receive standard surgery plus a saline (salt water) injection. During surgery, for patients in the treatment group, approximately 4mL (less than one teaspoon) of bone marrow will be taken from their hip bone using a special needle system. A small amount (1mL) will be sent to the laboratory for testing. Patients will be followed for 12 months after surgery and will complete questionnaires about their pain levels and knee function at several time points: before surgery, 2 weeks, 6 weeks, 3 months, 6 months, and 12 months after surgery. These questionnaires will ask about pain, daily activities, and overall improvement.

DETAILED DESCRIPTION:
There is a paucity of high-quality literature surrounding the efficacy of BMA in knee arthroscopy, and this study will help to fill this gap. The investigators can obtain preliminary data that indicates the effect of BMA on patient reported outcomes and also help identify evaluation end points for future BMA randomized trials. Additionally, this study will allow us to see how CFU, CD140, and CBC counts compare between BMA and BMAC. Our study will not be evaluating BMAC, just comparing the BMA numbers to previously reported BMAC counts. Cervos' BMA product could offer improved patient reported outcomes from knee arthroscopy. If this is true, this study could expand the reach of Cervos' BMA, improving the field of knee arthroscopy surgery and helping push orthopedics forward. Additionally, it could save surgeons and lab technicians time, and hospital's money, by removing the centrifugation step required in bone marrow concentrate products. Alternatively, no effect could help save patients money and help surgeons avoid this unnecessary treatment.

A total of 50 patients with osteoarthritis of the knee will be randomly assigned to receive arthroscopic debridement surgery or arthroscopic debridement surgery supplemented with bone marrow aspirate (BMA). Approximately 4mL of BMA will be obtained from different areas of the ilium using the Marrow Cellution™ aspiration system (Ranfac Corp., Avon, MA) following the manufacturer's instructions (Ranfac Technique Guide) intraoperatively for the patients in the treatment group. 1 mL of this will be set aside and sent to the lab for CBC, CD140 and CFU counts for comparison with other bone marrow aspirate products. Patients were randomized in equal numbers into either the treatment or control group (25 in each group). Patients and assessors of outcome were blinded to the treatment-group assignment. Outcomes were assessed at multiple points over a 12-month period with the use of five self-reported scores--three on scales for pain and two on scales for function--and one objective test of walking and stair climbing. The following measures will be included: IKDC, VAS, WOMAC, MARX, and PGIC will be collected at time points of baseline, 2 weeks, 6 weeks, and 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Require a primary knee arthroscopy for a meniscal injury or focal chondral defect (knee debridement or meniscectomy)
2. Have Kellgren-Lawrence grade 0 arthritis
3. Have Outerbridge cartilage grade 2 or lower
4. Ages 18-64

Exclusion Criteria:

1. Have previously undergone ipsilateral knee surgery
2. Have Kellegren-Lawrence grade 3 or greater
3. Have received other OrthoBiologics within 3 mo of surgery
4. Have ligament deficiencies
5. Need meniscal repair
6. Need a concomitant osteotomy or other realignment surgery
7. Have used DMARDs within the last three months
8. Have a hx of anemia, bleeding disorders, or inflammatory joint disease (rheumatoid arthritis, infectious arthritis, hemophilic arthropathy, Charcot's knee)
9. Have a hx of metabolic bone disease (osteoporosis, osteomalacia, rickets, osteitis fibrosa cystica, Paget's disease of bone)
10. Patients who are currently pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant patients are excluded from this study.
Enrollment: 50 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 12 month follow-up
  Knee Injury and Osteoarthritis Outcomes Score (KOOS)
  0-100 score range, with 0 representing extreme knee problems and 100 representing no knee problems.

CONTACTS AND LOCATIONS:
Overall Officials: Anil S Ranawat, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States